CLINICAL TRIAL: NCT00869414
Title: Comparison of Glycemic Response to Morning Only, Evening Only or Twice Daily Insulin Glargine in Patients With Type 1 Diabetes Using Continuous Glucose Monitoring
Brief Title: Glycemic Effects of Morning Only, Evening Only or Twice Daily Insulin Glargine in Patients With Type 1 Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI deceased
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00024168
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Results first posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-05

CONDITIONS: Type 1 Diabetes; Hypoglycemia
Keywords: hypoglycemia; type 1 diabetes; split dosing insulin glargine; continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Insulin Glargine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- insulin glargine only in morning (Active Comparator): Morning only administration of insulin glargine
  Interventions: Drug: Morning only administration of insulin glargine
- insulin glargine only at evening (Active Comparator): Evening only administration of insulin glargine
  Interventions: Drug: Evening only administration of insulin glargine
- split dose insulin glargine (Active Comparator): Split dose administration of insulin glargine, half dose in morning, half dose in evening
  Interventions: Drug: split dose insulin glargine

INTERVENTIONS:
Drug: Evening only administration of insulin glargine — Evening only administration of insulin glargine, with normal saline injection administered in the morning.
  Other Names: Lantus
  Arms: insulin glargine only at evening
Drug: Morning only administration of insulin glargine — Morning only administration of insulin glargine, with normal saline injection administered at night.
  Other Names: Lantus
  Arms: insulin glargine only in morning
Drug: split dose insulin glargine — split dose of insulin glargine, half administered in the morning, half administered in evening
  Other Names: Lantus
  Arms: split dose insulin glargine

SUMMARY:
This research is a prospective, randomized, cross-over study that is being done to compare the effect of morning only, evening only and twice daily insulin glargine (Lantus®) on hypoglycemia (blood glucose level <70 mg/dL) as measured by continuous glucose monitoring (CGM) in patients with type 1 diabetes.

DETAILED DESCRIPTION:
Over the course of the 6 week study, patients will take insulin glargine in each of 3 different times: only in the morning, only at night, and half in the morning, half at night. After 2 weeks taking the insulin in one regimen, patients will be switched to another regimen. Through the whole study, patients will be injecting themselves twice daily, and neither the patient nor the treating doctor will know which vials contain the insulin and which have only saline (placebo). The vials will be labeled MORNING or EVENING. Patients will continue to take their mealtime, short acting insulin doses.

Additionally, patients will wear a continuous glucose monitor (CGM) which will be masked. Before the study, patients will be taught about how to use the CGM, and keep it taped to their abdomen. The site that the CGM inserts into their abdomen will need to be changed every 5 days. We will know if a patients' blood sugar goes low even if the patient did not feel the low. Patients will still have to self-monitor their blood sugar levels at-least four times in five days, to calibrate the CGM.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women above age 18 with a diagnosis of type 1 diabetes mellitus
* On multiple insulin injections, including a long acting or intermediate acting insulin preparation and mealtime short acting insulin preparation.
* Clinical history consistent with hypoglycemia
* Hba1c <9.0%

Exclusion Criteria:

* Patients with type 2 diabetes mellitus
* Patients on insulin pump
* Poor control of diabetes (HbA1c > 9.0%)
* Pregnancy (women of childbearing age will undergo a pregnancy test at the start of the study and will be advised to use birth control methods during the study). Insulin glargine has been reported to have teratogenic effects in animal models, and therefore should only be used during pregnancy if clearly needed.
* Serious co-morbidities that, in clinical opinion of the investigators, could affect pharmacokinetics of glargine (e.g., CRF) or safety (e.g., recent CAD)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Saudek, MD, Principal Investigator — Johns Hopkins University; Ari S Eckman, MD, Study Director — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Garg SK, Gottlieb PA, Hisatomi ME, D'Souza A, Walker AJ, Izuora KE, Chase HP. Improved glycemic control without an increase in severe hypoglycemic episodes in intensively treated patients with type 1 diabetes receiving morning, evening, or split dose insulin glargine. Diabetes Res Clin Pract. 2004 Oct;66(1):49-56. doi: 10.1016/j.diabres.2004.02.008. PMID 15364161
- [Background] Ashwell SG, Gebbie J, Home PD. Twice-daily compared with once-daily insulin glargine in people with Type 1 diabetes using meal-time insulin aspart. Diabet Med. 2006 Aug;23(8):879-86. doi: 10.1111/j.1464-5491.2006.01913.x. PMID 16911626

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was prematurely terminated because the P.I. is deceased. Although 16 participants were enrolled, however, the number of participants starting and completing the study as well as the number of participants assigned to each Arm/Group are unknown, since no data are available
Period: Overall Study
Arm/Group | Insulin Glargine Only in Morning | Insulin Glargine Only at Evening | Split Dose Insulin Glargine
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This study was prematurely terminated because the PI is deceased. The Baseline data for the specific arms is unknown since no data are available. Only the baseline data for the overall population is available and reported.
Groups:
- All Study Participants: Participants were randomized to receive one of the three interventions: Insulin glargine only in the morning, Insulin glargine only in the evening, or a split dose of insulin glargine (half the dose in the morning and the other half in the evening).
Arm/Group | All Study Participants
Number analyzed (Participants) | 16
Age, Customized [Count of Participants; unit: Participants]
  Age, > 18 years old | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Time Spent (Mean Number of Minutes Per 24 Hour Day) in Hypoglycemic Range (<70mg/dl)
Time Frame: 6 weeks
Population: This study was prematurely terminated because the P.I. is deceased. The data for the Outcome Measures (if collected) is unknown since no data are available.
Arm/Group | Insulin Glargine Only in Morning | Insulin Glargine Only at Evening | Split Dose Insulin Glargine
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Change in the Mean Minutes Per 24 Hour Day in the Hyperglycemic Range of > 180 mg/dL.
Time Frame: 6 weeks
Population: as for outcome 1
Arm/Group | Insulin Glargine Only in Morning | Insulin Glargine Only at Evening | Split Dose Insulin Glargine
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: This study was prematurely terminated because the P.I. is deceased. The time frame for Adverse Event data (if collected) is unknown since no data are available.
Description: This study was prematurely terminated because the P.I. is deceased. The data for the Adverse Events (if collected) is unknown since no data are available.
Arm/Group | Insulin Glargine Only in Morning | Insulin Glargine Only at Evening | Split Dose Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes